CLINICAL TRIAL: NCT05859412
Title: Mechanisms of Neurodynamic Treatments (MONET)
Brief Title: Mechanisms of Neurodynamic Treatments
Acronym: MONET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Principal Investigator, ProfessorAnninaSchmid, A/Prof, PhD, MMACP, University of Oxford
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 313200
Record Dates: First submitted 2023-04-20; First posted 2023-05-16 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Carpal Tunnel Syndrome; Neurodynamic Treatment; Nerve Mobilisation; Diffusion MRI; Physiotherapy; Mechanistic Trial
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Steroids; Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor and the person responsible for the statistical analysis will be blinded to the participants' allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neurodynamic exercises (Experimental): 6-weeks home exercise programme of nerve and tendon gliding exercises
  Interventions: Other: Neurodynamic exercises
- Steroid injection Steroid injection (Depomedrone 40mg) (Active Comparator): Single steroid injection into Carpal Tunnel (positive control group)
  Interventions: Drug: Steroid injection (Depomedrone 40mg)
- Advice (Other): The advice group will receive advice but no additional intervention during the 6 week intervention period (negative control group)
  Interventions: Other: Advice

INTERVENTIONS:
Other: Neurodynamic exercises — The neurodynamic exercises will consist of a home-based exercise programme performed over a period of 6 weeks. Patients will attend a single session with an investigator who will instruct them the home exercise programme consisting of nerve and tendon gliding exercises which will be adjusted with pre-specified progressions over the 6 weeks intervention period. Patients will receive a leaflet and a video link detailing these exercises.
  Arms: Neurodynamic exercises
Drug: Steroid injection (Depomedrone 40mg) — Steroid injection (Depomedrone 40mg) into the carpal tunnel as per standard practice in patients with carpal tunnel syndrome
  Arms: Steroid injection Steroid injection (Depomedrone 40mg)
Other: Advice — Group receiving advice but no additional treatment
  Arms: Advice

SUMMARY:
INTRODUCTION: Carpal tunnel syndrome (CTS) is a relatively common condition caused by compression of one of the main nerves at the wrist, the median nerve. Non-surgical treatments, like steroid injections and physiotherapy, are the first line of treatment for patients with carpal tunnel syndrome. The investigators have previously shown that specific physiotherapeutic exercises (neurodynamic exercises) can reduce the need for carpal tunnel surgery in some patients. Experimental studies in animal models demonstrate that these exercises have an anti-inflammatory effect and can help the nerve to regenerate. However, the exact mechanisms of action of these exercises are not well understood in patients. A better understanding of the mechanisms of action of physiotherapeutic exercises would help clinicians to better target these treatments to those patients who may benefit from them.

AIM: To investigate the mechanisms of action of 6 weeks' neurodynamic treatments on nerve function and structure as well as patient-reported outcome measures in patients with CTS compared to a positive control intervention (routine care steroid injection) and a negative control intervention (advice).

METHODS AND ANALYSIS: In this single-blind randomised mechanistic trial, patients with confirmed mild to moderate CTS (n=78) and age and gender-matched healthy controls (n=30) will be included. Patients will be randomly allocated to a 6-week neurodynamic exercise group, steroid injection, or advice group. Outcome measures will be explored at baseline (patients and controls), post-intervention (patients), and 6-month follow-up (patients). Outcomes include diffusion-weighted and anatomical MRI of the median nerve at the wrist, quantitative sensory testing, nerve conduction studies, inflammatory markers in blood and skin biopsies, and validated questionnaires for pain, function, and psychological factors. Two-way repeated measures ANCOVAs (factors time and intervention, adjusted for baseline measurements as a continuous covariate) will be performed to identify differences in MRI parameters, clinical assessment, and inflammatory markers between patients in different groups and healthy controls.

DETAILED DESCRIPTION:
Follow-up at 6 months will only include outcome measures from questionnaires.

Details on enrollment:

Pilot testing of healthy participants who consented to our ethics but will not be included in the study was on 13-April-2023.

* First healthy participant enrolled: 17-May-2023.
* First patient participant enrolled: 1-June-2023.

Details on amendment:

* Amendment SA2_BPOR on 3/Aug/2023 to expand recruitment through registries of patients
* Amendment SA3_REC on 22/Aug/2023 to add Thames Valley Primary Care Research Partnership, musculoskeletal clinics, and media advertisement to help with recruitment of participants.

ELIGIBILITY:
Inclusion Criteria

Patients:

1. Patients who have a diagnosis of mild to moderate carpal tunnel syndrome based on a clinical assessment and confirmed with nerve conduction studies.
2. Male or Female, aged 18 years or above.
3. Patient is willing and able to give informed consent for participation in the study.

Healthy participants:

1. Male or female aged 18 years or above.
2. Participant is willing and able to give informed consent for participation in the study.
3. No history of hand or arm symptoms
4. No history of neck pain in the past 3 months
5. No systemic medical condition
6. No strong anticoagulant medication or altered coagulation (e.g., hemophilia) preventing skin biopsies
7. Severe anxiety or depression
8. Participants are required to be age- & sex-matched to patient participants
9. No contraindications for magnetic resonance scanning at 3T
10. Sufficient command of the English language

Exclusion Criteria

Patients:

1. Patients who already had surgery for their carpal tunnel syndrome (CTS) or are planning to undergo surgery in the next 6 weeks (patients with unilateral surgery who have unoperated CTS on the other hand are eligible to participate)
2. Patients who had a steroid injection for their CTS in the 6 months prior to the study enrolment or who had already more than 1 steroid injection into the study wrist.
3. Patients who have a diagnosis of severe carpal tunnel syndrome based on a clinical assessment and confirmed with electrodiagnostic testing
4. Electrodiagnostic testing revealing abnormalities other than CTS
5. Any other upper limb or neck problem for which they have sought treatment in the past 3 months
6. History of significant trauma to the upper limb or neck
7. Diabetes
8. Hypothyroidism
9. Severe anxiety or depression
10. Patient who is pregnant, lactating, or planning pregnancy during the study.
11. Patients on strong anticoagulant medication or altered coagulation preventing skin biopsies.
12. Contraindications for magnetic resonance imaging (assessed with MRI safety screening questionnaire).
13. Contraindications for steroid injections
14. Insufficient command of the English language

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-05-17 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Median nerve fractional anisotropy as determined on diffusion weighted imaging | Baseline
  Fractional anisotropy will be extracted from regions-of-interest in the median nerve and compared to healthy control group
Change in median nerve fractional anisotropy as determined on diffusion weighted imaging | From baseline to post-intervention (after 6-weeks)
  Change in fractional anisotropy extracted from regions-of-interest in the median nerve at post-intervention (after 6-weeks) compared to baseline

SECONDARY OUTCOMES:
Nerve markers on diffusion weighted imaging: water diffusivity (mm2/s) | Baseline
  Measured at the median nerve and cervical dorsal root ganglia. mm2/s; continuous data
Change to nerve markers on diffusion weighted imaging: water diffusivity (mm2/s) | From baseline to post-intervention (after 6-weeks)
  Measured at the median nerve and cervical dorsal root ganglia. mm2/s; continuous data
Nerve markers on anatomical MRI | Baseline
  Measured at the median nerve and cervical dorsal root ganglia. ratio/mm2; continuous data
Change in nerve markers on anatomical MRI | From baseline to post-intervention (after 6-weeks)
  Measured at the median nerve and cervical dorsal root ganglia. ratio/mm2; continuous data
Median nerve MRI T2 mapping | Baseline
  ms; continuous data
Changes in median nerve MRI T2 mapping | From baseline to post-intervention (after 6-weeks)
  ms; continuous data
Median nerve MRI magnetisation transfer ratio (MTR) | Baseline
  ratio; continuous data
Changes in median nerve MRI magnetisation transfer ratio (MTR) | From baseline to post-intervention (after 6-weeks)
  ratio; continuous data
Changes in median nerve conduction velocities from electrodiagnostic studies (m/s) | From baseline to post-intervention (after 6-weeks)
  m/s; continuous data
Changes in median sensory nerve action potentials (SNAPs) and compound muscle action potentials (CMAPs): amplitudes (mV) | From baseline to post-intervention (after 6-weeks)
  mV; continuous data
Thermal detection thresholds as assessed in Quantitative Sensory testing - warm and cold detection threshold; thermal sensory limen | Baseline
  Thermal detection thresholds will be assessed using a thermode over the index finger (e.g., ventral aspect of the proximal phalanx of the index finger).
  Data is measured in degrees celsius (point at which cold or warm is detected)
Change in thermal detection thresholds as assessed in Quantitative Sensory testing- warm and cold detection threshold; thermal sensory limen | From baseline to post-intervention (after 6-weeks)
  Thermal detection thresholds will be assessed using a thermode over the index finger (e.g., ventral aspect of the proximal phalanx of the index finger).
  Data is measured in degrees celsius (point at which cold or warm is detected)
Thermal pain thresholds as assessed in Quantitative Sensory testing- warm and cold painful threshold | Baseline
  Pain thermal thresholds will be assessed using a thermode over the index finger (e.g., ventral aspect of the proximal phalanx of the index finger) and over the contralateral lower limb (tibial anterior).
  Data is measured in degrees celsius (point at which cold or warm is initially detected as painful)
Change in thermal pain thresholds as assessed in Quantitative Sensory testing- warm and cold painful threshold | From baseline to post-intervention (after 6-weeks)
  Pain thermal thresholds will be assessed using a thermode over the index finger (e.g., ventral aspect of the proximal phalanx of the index finger) and over the contralateral lower limb (tibial anterior).
  Data is measured in degrees celsius (point at which cold or warm is initially detected as painful)
Mechanical detection thresholds as assessed in Quantitative sensory testing | Baseline
  Mechanical detection thresholds will be assessed using a standardised set of von Frey filaments (mN) over the index finger. Geometric mean will be calculated
Change in mechanical detection thresholds as assessed in Quantitative sensory testing | From baseline to post-intervention (after 6-weeks)
  Mechanical detection thresholds will be assessed using a standardised set of von Frey filaments (mN) over the index finger. Geometric mean wil be calculated
Mechanical pain thresholds as assessed in Quantitative sensory testing | Baseline
  Mechanical pain thresholds will be assessed using a series of weighted pin prick stimulators (mN). They will be assessed over the index finger and over the contralateral lower limb (tibial anterior).
Change in mechanical pain thresholds as assessed in Quantitative sensory testing | From baseline to post-intervention (after 6-weeks)
  Mechanical pain thresholds will be assessed using a series of weighted pin prick stimulators (mN). They will be assessed over the index finger and over the contralateral lower limb (tibial anterior).
Mechanical pain sensitivity as assessed in Quantitative sensory testing | Baseline
  Mechanical pain sensitivity will be assessed using a series of weighted pin prick stimulators (mN) over the index finger. Pain rating for each stimulus on a 0-100 numerical rating scale ('0' indicating "no pain", and '100' indicating "most intense pain imaginable"). Geometric mean of all numerical ratings for pinprick stimuli will be calculated
Change in mechanical pain sensitivity as assessed in Quantitative sensory testing | From baseline to post-intervention (after 6-weeks)
  Mechanical pain sensitivity will be assessed using a series of weighted pin prick stimulators (mN) over the index finger. Pain rating for each stimulus on a 0-100 numerical rating scale ('0' indicating "no pain", and '100' indicating "most intense pain imaginable"). Geometric mean of all numerical ratings for pinprick stimuli will be calculated
Dynamic mechanical allodynia as assessed in Quantitative sensory testing | Baseline
  Pain rating for each stimulus on a 0-100 numerical rating scale ('0' indicating "no pain", and '100' indicating "most intense pain imaginable"). Geometric mean (compound measure) of all numerical ratings across light touch stimulators over the index finger
Change in dynamic mechanical allodynia as assessed in Quantitative sensory testing | From baseline to post-intervention (after 6-weeks)
  Pain rating for each stimulus on a 0-100 numerical rating scale ('0' indicating "no pain", and '100' indicating "most intense pain imaginable"). Geometric mean (compound measure) of all numerical ratings across light touch stimulators over the index finger
Wind-up ratio as assessed in Quantitative sensory testing | Baseline
  Wind-up ration will be assessed using a pin prick (mN) over the index finger (e.g., ventral aspect of the proximal phalanx of the index finger). Ratio, continous data
Change in wind-up ratio as assessed in Quantitative sensory testing | From baseline to post-intervention (after 6-weeks)
  Change in wind-up ration will be assessed using a pin prick (mN) over the index finger (e.g., ventral aspect of the proximal phalanx of the index finger). Ratio, continuous data
Vibration detection thresholds as assessed in Quantitative sensory testing | Baseline
  Vibration detection thresholds will be assessed using a tuning fork (64 Hz, 8/8 scale) over a bony prominence over (e.g., palmar side of the distal end of the second metacarpal)
Change in vibration detection thresholds as assessed in Quantitative sensory testing | From baseline to post-intervention (after 6-weeks)
  Change in vibration detection thresholds will be assessed using a tuning fork (64 Hz, 8/8 scale) over a bony prominence over (e.g., palmar side of the distal end of the second metacarpal)
Pressure pain thresholds as assessed in Quantitative sensory testing | Baseline
  Pressure pain thresholds will be assessed using an algometer (kg) on the thenar eminence and over the contralateral lower limb (tibialis anterior)
Change in pressure pain thresholds as assessed in Quantitative sensory testing | From baseline to post-intervention (after 6-weeks)
  Change in pressure pain thresholds will be assessed using an algometer (kg) on the thenar eminence and over the contralateral lower limb (tibialis anterior)
Pinch strength test - maximum isometric strength | Baseline
  Pinch grip dynamometry. Continuous data, kg
Change in pinch strength test - maximum isometric strength | From baseline to post-intervention (after 6-weeks)
  Pinch grip dynamometry. Continuous data, kg
Nerve mechanosensitivity- upper limb neurodynamic test (median nerve) | Baseline
  Evaluation of nerve mechanosensitivity in response to mechanical load (increased tension) applied to the nerve. Range of elbow extension at point of symptoms (degrees)
Change in nerve mechanosensitivity- upper limb neurodynamic test (median nerve) | From baseline to post-intervention (after 6-weeks)
  Change in nerve mechanosensitivity in response to mechanical load (increased tension) applied to the nerve. Range of elbow extension at point of symptoms (degrees)
Nerve mechanosensitivity - positive upper limb neurodynamic tests | Baseline
  Upper limb neurodynamic tests will be assessed to determine the presence of increased mechanosensitivity. The neurodynamic test will be graded as 'positive', when there is at least partial reproduction of symptoms plus when symptoms can be modified with structural differentiation. Otherwise, the neurodynamic test will be graded as 'negative'
Change in nerve mechanosensitivity - positive upper limb neurodynamic tests | From baseline to post-intervention (after 6-weeks)
  Upper limb neurodynamic tests will be assessed to determine the presence of increased mechanosensitivity. The neurodynamic test will be graded as 'positive', when there is at least partial reproduction of symptoms and when symptoms can be modified with structural differentiation. Otherwise, the neurodynamic test will be graded as 'negative'
Symptom severity and limitations in hand function as assessed by the Boston carpal tunnel syndrome questionnaire | Baseline, post-intervention (after 6 weeks), 6-months follow up
  Patient reported symptoms and limitations on the Boston carpal tunnel syndrome questionnaire
Symptom intensity levels on a Visual Analogue Scale (VAS) | Baseline, post-intervention (after 6 weeks), 6-months follow up
  Patient reported average intensity of pain, paraesthesia and numbness on 10cm visual analogue scales, ranging from no symptoms to worst symptoms ever
Location of symptoms in a body and a hand diagram | Baseline, post-intervention (after 6 weeks)
  Patient reported location of symptoms in a body diagram and a hand diagram.
Presence of central sensitisation as assessed with the Central Sensitisation Inventory | Baseline, post-intervention (after 6 weeks), 6-months follow up
  Patient reported central sensitisation on the Central Sensitisation Inventory
Functional deficits- Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire | Baseline, post-intervention (after 6 weeks), 6-months follow up
  Participant reported outcomes on ability to perform activities as per quick DASH questionnaire
Functional deficits- Patient specific functional scale (PSFS) | Baseline, post-intervention (after 6 weeks), 6-months follow up
  Participant reported outcomes on the patient specific functional scale
Presence of neuropathic pain - DN4 | Baseline, post-intervention (after 6 weeks), 6-months follow up
  Patient screened for neuropathic pain using DN4
Presence of neuropathic pain - pain DETECT | Baseline, post-intervention (after 6 weeks), 6-months follow up
  Patient screened for neuropathic pain using pain DETECT
Neuropathic pain symptoms - Neuropathic Pain Symptom Inventory | Baseline, post-intervention (after 6 weeks), 6-months follow up
  Patient reported outcomes on neuropathic pain symptoms as assessed on Neuropathic Pain Symptom Inventory.
Presence of psychological co-morbidities - The Depression, Anxiety, and Positive Outlook Scale (DAPOS) | Baseline, post-intervention (after 6 weeks), 6-months follow up
  Participant reported outcomes on depression and anxiety as per DAPOS
Presence of psychological co-morbidities - short-form Pain Anxiety Symptoms Scale (PASS-20) | Baseline, post-intervention (after 6 weeks), 6-months follow up
  Participant reported outcomes on depression and anxiety as per short-form Pain Anxiety Symptoms Scale (PASS-20)
Presence of psychological co-morbidities - pain catastrophizing scale (PCS) | Baseline, post-intervention (after 6 weeks), 6-months follow up
  Participant reported outcomes on depression and anxiety as per pain catastrophising scale (PCS)
Assessment of quality of life - EQ-5D-5L | Baseline, post-intervention (after 6 weeks), 6-months follow up
  Participant reported outcomes on quality of life as per EQ-5D-5L questionnaire
Assessment of sleep interference - Insomnia Severity Index | Baseline, post-intervention (after 6 weeks), 6-months follow up
  Participant reported outcomes on sleep interference with the Insomnia Severity Index.
Adverse and serious adverse events | From start of intervention until end of intervention (6 weeks)
  Patient self-reported adverse events
Exercise adherence to the neurodynamic home-based intervention - number of sessions | From start of intervention until end of intervention (6 weeks)
  Patient self-reported number of sessions per day throughout the intervention in an exercise diary

OTHER OUTCOMES:
Blood samples - DNA | Baseline
  Blood samples coupled with detailed phenotype data will investigate potential gene associations in CTS and recovery
Change in blood samples - DNA | From baseline to post-intervention (after 6-weeks)
  Change in blood samples coupled with detailed phenotype data will investigate potential gene associations in CTS and recovery
Concentration of serum inflammatory markers - metabolomics | Baseline
  Concentrations of inflammatory markers in serum
Change in the concentration of serum inflammatory markers - metabolomics | From baseline to post-intervention (after 6-weeks)
  Change in the concentrations of inflammatory markers in serum
Pro-inflammatory cytokine levels | Baseline
  Proinflammatory cytokine assay (pg/ml); continuous data
Change in pro-inflammatory cytokine levels | From baseline to post-intervention (after 6-weeks)
  Change in proinflammatory cytokine assay (pg/ml); continuous data
Concentration of inflammatory markers in serial skin biopsies | Baseline
  Concentration of inflammatory markers in skin biopsies. Baseline biopsy will be performed in the most distal part of the ventrolateral side of the proximal phalanx of the index finger. The 6-weeks biopsy will be performed proximally, avoiding the primary biopsy site
Change in concentration of inflammatory markers in serial skin biopsies | From baseline to post-intervention (after 6-weeks)
  Change in concentration of inflammatory markers in skin biopsies. Baseline biopsy will be performed in the most distal part of the ventrolateral side of the proximal phalanx of the index finger. The 6-weeks biopsy will be performed proximally, avoiding the primary biopsy site

CONTACTS AND LOCATIONS:
Overall Officials: Eva Sierra-Silvestre, PhD, Principal Investigator — University of Oxford
Locations (1):
- Nuffield Department of Clinical Neurosciences, University of Oxford, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All IPDs that underlie results in a publication.
Supporting Information: Study Protocol
Time Frame: IPD that underlie results of a publication will be shared upon the final publication of the main manuscripts of this study.
Access Criteria: IPD will be shared upon reasonable request and in line with ethical approval with authors contacting the study investigators.

REFERENCES:
- [Derived] E SS, M T, Ac T, M S, G B, Ab S. Mechanisms of neurodynamic treatments (MONET): a protocol for a mechanistic, randomised, single-blind controlled trial in patients with carpal tunnel syndrome. BMC Musculoskelet Disord. 2024 Jul 27;25(1):590. doi: 10.1186/s12891-024-07713-6. PMID 39068435